CLINICAL TRIAL: NCT02860416
Title: Additional Post Hoc Analysis and Clinical Data Collection for Subjects Tested With Brain Network Activation (BNA™) Technology
Brief Title: Additional Post Hoc Analysis and Clinical Data Collection
Acronym: BNA™
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-28
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Neurological Observations
Keywords: Neurology
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect additional Investigational cognitive tasks and additional clinical data for subjects tested with ElMindA's Brain Network Activation (BNA™).

DETAILED DESCRIPTION:
To collect additional Investigational cognitive tasks and additional clinical data for subjects tested with ElMindA's Brain Network Activation (BNA™).

The BNA™ technology was developed and is utilized by ElMindA Ltd. The (BNA™) Analysis System is cleared for use by qualified medical professionals for the post hoc statistical analysis of the human electroencephalogram ("EEG"), utilizing evoked response potentials ("ERP').

ELIGIBILITY:
Inclusion Criteria:

* Completed a BNA test in the past
* Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments.
* Willingness to participate

Exclusion Criteria:

* Significant Sensory deficit

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who completed a BNA test with the Auditory Oddball Task, from both genders, aged 3-99 years.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-07; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
engineering development according to clinical assessments | 2 years
  The study is designed to collect data that will aid in future scientific and engineering exploration of correlations between clinical assessments and BNA scores. The results are primarily intended for scientific inquiry and engineering development purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Skopin, PhD, Principal Investigator — ElMindA Ltd
Locations (2):
- United States (2):
  - ElMindA, Glenview, Illinois
  - Premier Psychiatric Group, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No